CLINICAL TRIAL: NCT01919385
Title: Feasibility Study Assessing the Ability of an Insulin Pump-controlling Algorithm to Minimize Hypoglycemia in Patients With Type 1 Diabetes in a Clinical Research Setting
Brief Title: Feasibility Study Assessing the Ability of an Insulin Pump-controlling Algorithm to Minimize Hypoglycemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Animas Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3108873,
Record Dates: First submitted 2013-06-28; First posted 2013-08-09 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- type 1 diabetes (Experimental): Predictive Low Glucose Minimizer (PLGM) System
  Interventions: Device: Predictive Low Glucose Minimizer

INTERVENTIONS:
Device: Predictive Low Glucose Minimizer — This study is a non-randomized feasibility study enrolling type 1 diabetics who are currently using an insulin pump. Participating Investigators will closely monitor the study subject in a clinical research center environment for approximately 30 hours, while controller algorithm determined insulin doses are delivered by an insulin pump, and utilizing continuous glucose monitoring results.
  Other Names: type 1 diabetes

SUMMARY:
This study will be conducted in a Clinical Research Center (CRC) setting and recruiting type 1 diabetes that are currently using an insulin pump.

DETAILED DESCRIPTION:
This study is a non-randomized, uncontrolled feasibility study that looks to enroll people with type 1 diabetes who are currently using an insulin pump. During the subject's participation, the study staff will closely monitor the study subject in a clinical research center environment for approximately 30 hours, while controller algorithm determined insulin doses are delivered by an insulin pump, and utilizing continuous glucose monitoring results.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65 years
* Type 1 diabetes mellitus for at least one year
* Currently using an insulin infusion pump for at least the past 6 months

Exclusion Criteria:

* Pregnancy
* History of Diabetic Ketoacidosis (DKA) in the past six months
* History of severe hypoglycemia (Seizure, unconsciousness) in the past 6 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance of the System while the subject is under close medical supervision in the Clinical Research Center (CRC) setting | 1 week after subject is enrolled in the study
  Evaluating the ability of the system to predict a fall or rise in glucose values below or above a low glucose threshold, and take the corresponding appropriate action of reducing or suspending insulin delivery in order to keep the subject's glucose above this threshold, or resuming insulin delivery at the current basal rate upon the increase of glucose above this threshold.
  Ability of the system to issue timely and accurate warnings.

SECONDARY OUTCOMES:
Capturing the number of Adverse Events as a measure of assessing subject safety | 1 week after subject is enrolled in the study
  Understand the System's ability to safely keep the subject glucose levels within designated threshold. The subject and the device will be continuously monitored by the Principle Investigator and Algorithm Engineer to ensure proper function of the device and subject safety. All Adverse Events will be captured on the CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Zisser, MD, Principal Investigator — Samsum Diabetes Reserach Inst.
Locations (1):
- Samsum Diabetes Reserach Inst., Santa Barbara, California, United States

REFERENCES:
- [Derived] Finan DA, Dassau E, Breton MD, Patek SD, McCann TW Jr, Kovatchev BP, Doyle FJ 3rd, Levy BL, Venugopalan R. Sensitivity of the Predictive Hypoglycemia Minimizer System to the Algorithm Aggressiveness Factor. J Diabetes Sci Technol. 2015 Jun 30;10(1):104-10. doi: 10.1177/1932296815593292. PMID 26134834